CLINICAL TRIAL: NCT01280019
Title: Functional Residual Capacity Guided Alveolar Recruitment Strategy in Patients With Acute Respiratory Failure After Cardiac Surgery
Brief Title: FRC Guided Therapy in Acute Respiratory Failure
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Luebeck (Other)
Collaborators: European Society of Intensive Care Medicine (Other)
Responsible Party: Dr. Hermann Heinze, Department of Anaesthesiology, University of Lübeck
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FRC-ARF
Record Dates: First submitted 2011-01-19; First posted 2011-01-20 (Estimated); Last update posted 2011-01-20 (Estimated); Status verified 2011-01

CONDITIONS: Mechanical Ventilation; Acute Respiratory Failure; Cardiac Surgery
Keywords: functional residual capacity; electrical impedance tomography; inflammatory parameters

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- FRC guided (Experimental): Patients receive an alveolar recruitment manoeuvre if FRC falls below 94% of baseline FRC
  Interventions: Procedure: alveolar recruitment manoeuvre
- Saturation guided (Active Comparator): Patients receive an alveolar recruitment manoeuvre if peripheral oxygen saturation falls below 90%
  Interventions: Procedure: alveolar recruitment manoeuvre

INTERVENTIONS:
Procedure: alveolar recruitment manoeuvre — Increase of airway pressures in a stepwise manner from set peak inspiratory pressure/ positive end-expiratory pressure up to 40/15 mbar and back over 2 minutes.

SUMMARY:
In ventilated patients with acute respiratory failure endotracheal suctioning may lead to alveolar derecruitment, which can be monitored by means of functional residual capacity (FRC) measurements. Regional distribution of ventilation can be followed at bedside using electrical impedance tomography. The investigators hypothesize that a FRC guided recruitment strategy, aimed at restoring a baseline FRC value after open endotracheal suctioning, improves oxygenation and regional distribution of ventilation. In addition the investigators research the impact of such a strategy on the inflammatory response to mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* need for mechanical ventilation due to respiratory failure after cardiac surgery

Exclusion Criteria:

* circulatory failure, eg. need for high doses of inotropes or extracorporal cardiac support

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-12 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Regional ventilation | 6 hours
  Regional distribution of ventilation over 6 hours of treatment

SECONDARY OUTCOMES:
arterial oxygenation and inflammation | 6 hours
  Changes of arterial oxygenation and inflammatory parameters in the blood during 6 hours of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesiology, Intensive Care Unit, University of Lübeck, Lübeck, Germany